CLINICAL TRIAL: NCT06366035
Title: Leveraging on Virtual Engagement for Maternal Understanding & Mood-enhancement "LoVE4MUM" Mobile Application- A Protocol for Pilot Randomized Control Trial for Preventing Postpartum Depression
Brief Title: LoVE4MUM: Virtual Engagement for Preventing Postpartum Depression
Acronym: LoVE4MUM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Institutes of Health, Ministry of Health Malaysia (Other)
Responsible Party: Principal Investigator, Siti Sabrina binti Kamarudin, Principal Investigator, National Institutes of Health, Ministry of Health Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NMRR ID-24-00924-HPO
Record Dates: First submitted 2024-04-10; First posted 2024-04-15 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Postpartum Depression; Maternal Behavior; mHealth Intervention; Mental Health Issue
Keywords: Postpartum Depression; mHealth intervention; self-guided; postpartum mental health literacy
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Intervention Model Description: Single Blinded, Pilot Randomized Control Trial
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as Usual (TAU) (No Intervention): Mothers receiving treatment as usual (TAU) at the postpartum health care facilities according to standard guideline from period of delivery up to 6 weeks postpartum
- Treatment as Usual & LoVE4MUM phone application (Experimental): Mothers receiving treatment as usual (TAU) and LoVE4MUM phone application from period of delivery up to 6 weeks postpartum
  Interventions: Device: LoVE4MUM mobile application

INTERVENTIONS:
Device: LoVE4MUM mobile application — LoVE4MUM is an innovative mobile application developed based on cognitive behavioral therapy and psychoeducation. The mobile application consist of 5 main modules which delivers information pertaining self-care, postpartum depression, handling negative thoughts, mood tracking and information for seeking help. The module consist of short notes, videos and worksheets for the participants to conduct.
  Arms: Treatment as Usual & LoVE4MUM phone application

SUMMARY:
Postpartum depression is a serious concern affecting mothers and their infants, especially with limited traditional support. This pilot study evaluates the effectiveness of a novel mobile app called LoVE4MUM, developed based on Cognitive Behavioral Therapy and Psychoeducation principles, in preventing postpartum depression. The pilot trial involves 64 mothers randomly assigned to receive either standard care or standard care plus the LoVE4MUM. Primary outcome is improvement in depression, with secondary outcomes including mental health literacy and automatic negative thoughts. This research aims to provide initial evidence on the potential of mobile health tools to support maternal mental health, paving the way for future accessible and effective interventions.

DETAILED DESCRIPTION:
Postpartum depression (PPD) is a significant mental health issue. Traditional support systems remains challenging and mHealth intervention provides an opportunity to access for support.

The primary objective of this study is to preliminarily assess the effectiveness of a developed mobile application called LoVE4MUM in prevention of postpartum depression. The study will employ a single-blinded, pilot randomized controlled trial (RCT) design involving a sample of 64 mothers. Participants will be randomly assigned in a 1:1 ratio to one of two groups: the intervention group, which will receive standard postpartum care plus LoVE4MUM mobile application, or the control group, which will receive standard postpartum care alone. The primary outcome measure will be the effectiveness of the mobile application in improving symptoms of postpartum depression among mothers. Secondary outcome measures will include changes in postpartum mental health literacy scores and negative automatic thoughts frequencies.

Through the systematic evaluation of the LoVE4MUM mobile application in conjunction with standard postpartum care, this pilot RCT aims to generate preliminary evidence regarding the efficacy and feasibility of using mHealth tools for preventing postpartum depression.

ELIGIBILITY:
Inclusion Criteria:

* mothers with EPDS score 9-<12
* mothers with access to smartphone and internet connectivity
* continue routine postpartum care at the government health facilities
* literate in english and malay

Exclusion Criteria:

* history of drug abuse
* diagnosis of depressive illness or any other mental health illness
* undergoing treatment for mental health
* infant born with intrauterine death or died immediately after birth

Ages: 19 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-04-22 (Estimated); Primary Completion 2024-06-03 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Postpartum Depression | Baseline, 1 week and 6 weeks postpartum
  Self report measure using the Edinburgh Postpartum Depression Scale (EPDS) by the subjects on their symptoms of emotional distress during pregnancy and the postnatal period. Scale has been validated in English and Malay language with a total of 10 items based on 4 point Likert scale (0-3). Expected scoring 0 - 30. Score above 12 is considered probable depression.

SECONDARY OUTCOMES:
Postpartum Mental Health Literacy | Baseline, 1 week and 6 weeks postpartum
  self report measure using the Postpartum Depression Literacy Scale (PoDLiS) by the subjects on their knowledge and attitude on postpartum depression, help seeking, symptoms and available support. It has been validated in English and the Malay language. The 31 items is rated on a 5 point Likert scale (1-5). Total score is the total raw score divided by the total item. Higher score equivalents to higher postpartum mental health literacy
Automatic Negative Frequency | Baseline, 1 week and 6 weeks postpartum
  self report measure using the Automatic Thoughts Questionnaire (ATQ) by the subjects on the frequency of experiencing the negative thought statement. It has been validated in the English and Malay language. The 17 items is rated based on a 5 point Likert scale (1-5). Total score 17- 85. Higher score equivalent to higher frequency of negative thoughts.

CONTACTS AND LOCATIONS:
Overall Officials: Siti Sabrina Kamarudin, MBBS, Principal Investigator — National Institute for Health, NIH Malaysia
Locations (2):
- Malaysia (2):
  - Hospital Tengku Ampuan Rahimah, Klang, Selangor
  - Hospital Shah Alam, Shah Alam, Selangor

IPD SHARING:
Plan to Share IPD: No
information could be available upon reaching out to the principal investigator. However date relative to the time when summary data are published or otherwise made available starting 6 months after publication.

REFERENCES:
- [Derived] Kamarudin SS, Idris IB, Sharip S, Ahmad N. LoVE4MUM Mobile App to Prevent Postpartum Depression: Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2025 Jan 27;14:e63564. doi: 10.2196/63564. PMID 39869891